CLINICAL TRIAL: NCT00787904
Title: The Role of T-cells in Women Undergoing Surgical Menopause
Brief Title: Role of T-cells in Post-Menopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Associate Professor, Atlanta VA Medical Center
Other Study IDs: T-cells in osteoporosis
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, T-cells
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Surgical Menopause: Pre-menopausal women undergoing total hysterectomy with oophorectomy rendering them post-menopausal
- Surgical Control: Pre-menopausal women undergoing abdominal surgery but without ovary removal
- Healthy: Healthy matched pre-menopausal controls

SUMMARY:
This is an observational study of women undergoing surgical menopause to determine whether T-cells play an important role in the etiology of post-menopausal osteoporosis. Subjects will examined before and after surgery and followed over a two year period to determine the biology of T-cells during this study period.

DETAILED DESCRIPTION:
Estrogen (E) deficiency is a major cause of post-menopausal osteoporosis. The mechanisms by which E deficiency causes osteoporosis has been recently linked to regulation of two key osteoclastic cytokines: RANKL and TNFα (TNF) , , produced by the T-cell in the bone micro-environment. TNF is a cytokine that has long been associated with bone destruction during E deficiency in both animal and human models. However, the cellular sources of TNF and its exact mechanism of action are poorly understood. Previous studies in animal models has demonstrated that in marked contrast to responses in wild type (WT) mice, ovariectomy (ovx) failed to induce bone loss and did not stimulate osteoclast (OC) formation in T-cell deficient mice. This phenomenon is reversed by T cell reconstitution with WT T cells but not with T cells from TNF -/- mice2,4. These findings established T-cells and T-cell produced TNF as essential mediators of the bone-wasting effects of E deficiency in vivo. TNF further enhances OC formation by up regulating the stromal cell production of RANKL and M-CSF and by augmenting the responsiveness of OC precursors to RANKL4. The mechanisms by which E deficiency leads to enhanced levels of T-cell derived TNF involve a realignment of the adaptive immune response that ultimately leads to an expansion in the pool of TNF secreting T-cells. Dr. Pacifici's group showed that these pathways in mouse models involve the up-regulation of antigen presentation by macrophages and dendritic cells, leading to T cell activation and peripheral expansion of TNF producing T cells. They also showed that E deficiency causes a rebound in thymic T cell output that contributes to both the T cell expansion and the bone loss induced by ovx in young adult mice .

The objective of this study is to translate these critical findings in the mouse for the first time to E deficient women following ovx. If this work defines an important role for T-cells in E deficiency-induced bone loss, this could stimulate the development of novel therapies designed to block T-cell expansion or their contribution to cytokine production and thus prevent or attenuate bone loss in this common clinical setting. The hypothesis of the research plan is that T-cells derived from women, rendered E deficient after undergoing ovx, exhibit: 1) increased T-cell activation, and proliferation; 2) enhanced production of pro-osteoclastogenic cytokines RANKL and TNF; and 3) demonstrate increased T-cell output from the thymus that together cause bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Women between the age of 18-55, pre-menopausal by history (regular spontaneous menstrual bleeding every 21-35 days) or documented FSH <10, no current estrogen therapy, undergoing hysterectomy with (ovx) or without ovariectomy (control group) for benign gynecologic disease (fibroid uterus, endometriosis, dysfunctional uterine bleeding, chronic pelvic pain) or for prophylaxis against ovarian cancer (BRCA positive).

Exclusion Criteria:

* History of an active cancer including breast and uterine cancer, treatment with chemotherapy or glucocorticoids
* History of an immune deficiency syndrome including HIV infection
* History of severe anemia with hematocrit < 25.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-menopausal Women
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, M.D./Ph.D., Principal Investigator — Emory University/Atlanta VAMC
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Control: Pre-menopausal women with or without surgery
Period: Overall Study
Arm/Group | Surgical Menopause | Surgical Control
Started | 6 | 13
Completed | 6 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Menopause | Surgical Control | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (5.1) | 41.4 (7.1) | 42.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in T-cell Activation Measured by Flow Cytometry, Specifically the Percentage of CD3+CD69+ T-cells
Description: (Please note to reviewer, CD3 positivity indicates a T-cell, the title is correct)
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: percentage of CD3 positive cells
Arm/Group | Surgical Menopause | Surgical Control
Number analyzed (Participants) | 6 | 13
percentage of CD3 positive cells | 3.6 (0.5) | 1.8 (0.2)

2. Primary Outcome: Percent Change in Thymus Size Measured by CT Scan
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Surgical Menopause | Surgical Control
Number analyzed (Participants) | 6 | 13
percent change | -7 (2) | 17 (4)

3. Secondary Outcome: Bone Mineral Density
Description: Please note that the bone density measurements were done AFTER THE PRIMARY endpoints because bone mineral density changes take longer to see differences
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Surgical Menopause | Surgical Control
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/13
Other Adverse Events (participants affected / at risk) | 0/6 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No